CLINICAL TRIAL: NCT03179917
Title: Pembrolizumab and Involved Site Radiation Therapy for Early Stage Relapsed or Primary Refractory Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-054
Record Dates: First submitted 2017-06-06; First posted 2017-06-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Hodgkin Lymphoma
Keywords: Pembrolizumab; Radiation Therapy; 17-054
MeSH Terms: conditions — Hodgkin Disease | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: This phase II study will use an optimal Simon two-stage design.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Involved Site Radiation Therapy (Experimental): Following a PET/CT simulation to evaluate the extent of disease, pembrolizumab 200mg IV will be given over 30 minutes on day 1 of each 21 day cycle for a total of 4 cycles. Fourteen to 21 days after the completion of therapy, a PET/CT simulation will be repeated. Pts with complete response will proceed to 20 Gy of ISRT. Pts without a PET CR, but improvement on CT scan will have a repeat biopsy. If the biopsy is negative for Hodgkin Lymphoma, these ps will receive 30 Gy of ISRT. If the biopsy is positive for Hodgkin Lymphoma, they will receive 36-40 Gy ISRT. Pts without a PET CR, but improvement on CT scan will have a repeat biopsy. If the biopsy is negative for Hodgkin Lymphoma, these pts will receive 30 Gy of ISRT. If the biopsy is positive for Hodgkin Lymphoma, they will receive 36-40 Gy ISRT. Pts with new sites of disease or progression on imaging will have a repeat biopsy, per treating physician's discretion & then be treated off study.
  Interventions: Drug: Pembrolizumab; Radiation: Involved Site Radiation Therapy

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab 200mg IV will be given over 30 minutes on day 1 of each 21 day cycle for a total of 4 cycles. Pediatric patients will be treated at 2 mg/kg with a maximum dose of 200 mg.
Radiation: Involved Site Radiation Therapy — 30 Gy of ISRT

SUMMARY:
This study is being done to test the safety and effectiveness of pembrolizumab followed by radiation therapy in Hodgkin lymphoma.

The purpose of this study is to determine how effective combining the research drug, pembrolizumab, with a targeted form of radiation therapy known as involved site radiotherapy can be in patients with relapsed or refractory early stage classical Hodgkin lymphoma. The goal is to see whether this treatment strategy can cure a significant number of patients with relapsed or refractory early stage classical Hodgkin lymphoma while avoiding the toxicity of either a large radiation field or further chemotherapy and stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Three populations of patients are eligible for enrollment:

  (1) Patients with early stage disease at diagnosis (stage I-II) who were treated with chemotherapy alone and relapsed with early stage disease (stage RI-II).

  (2) Patients with early stage disease at diagnosis (stage I-II) who were treated with chemotherapy alone and have early stage (stage RI-II) primary refractory disease (residual disease on a scan 1 month after the completion of initial therapy) without B-symptoms and with each area of disease less than 10 cm in size.

  (3) Patients with early stage disease at diagnosis (stage I-II) who were treated with combined modality therapy (chemotherapy and radiation) who relapse with early stage disease (stage RI-II) outside the prior radiation therapy field.
* Histologic confirmation of classical Hodgkin Lymphoma after imaging documenting primary refractory or relapsed disease
* Age 12 or older
* ECOG Performance Status of 0-1 or Lansky Performance Status of ≥ 50 (Pts 12-15 years of age)
* Adequate organ function. Screening labs should be performed within 14 days of treatment initiation.

Hematologic

* Absolute neutrophil count (ANC) ≥1,000 /mcL
* Platelets* ≥75,000 / mcL
* Hemoglobin* ≥8 g/dL Renal
* Creatinine OR Measured or calculated** creatinine clearance CrCl (GFR can also be used in place of creatinine or ≤1.5 X upper limit of normal for age (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN Hepatic
* Total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels >1.5 ULN
* AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for age for subjects with liver involvement Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy, then as long as PT or PTT is within therapeutic range of intended use of anticoagulants

  * 1.5 X ULN unless subject is receiving anticoagulant therapy, then as long as PT or PTT is within therapeutic range of intended use of anticoagulants * Hemoglobin and platelet requirements cannot be met by use of recent transfusion or growth factor support (GCSF or erythropoietin) within 2 weeks prior to treatment initiation.

    * Creatinine clearance should be calculated per institutional standard.

      * Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from sexual activity for the course of the study through 120 days after the last dose of study medication (Reference Section 5.7.2). Subjects of child bearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

Note: Abstinence is acceptable if this is the established and preferred contraception for the subject.

* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the established and preferred contraception for the subject.

Exclusion Criteria:

* Ann Arbor Stage III or IV disease at diagnosis or at relapse/refractory disease confirmation.
* Bulky disease (>10cm) at diagnosis or at relapse/refractory disease confirmation.
* Active B symptoms.
* Received >1 line of therapy for Hodgkin lymphoma
* Relapsed/refractory disease within a prior radiation field.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Diagnosis of immunosuppression or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has history of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non infectious pneumonitis
* Has an active infection requiring intravenous systemic therapy.
* Has a known Human Immunodeficiency Virus (HIV), Hepatitis B (HBV), or Hepatitis C (HCV) infection
* Has received a live vaccine or live attenuated vaccine within 30 days prior to first dose of study drug. Administration of killed vaccines is allowed
* Any other medical condition or laboratory evaluation that, in the treating physician's or principal investigator's opinion, makes the patient unsuitable to participate in this clinical trial
* Has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e. ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has had treatment a prior monoclonal antibody targeting PD-1, PD-L1, PD-L2, or CTLA-4.
* Has a pre-treatment TTE showing a calculated left ventricular ejection fraction of less than 50%
* Has a pre-treatment PFT showing an DLCO adjusted for hemoglobin of less than 60%
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-06-08 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
complete response rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - University of Miami, Miami, Florida
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Abramson Cancer Center at University of Pennsylvania (Data Collection Only), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm